CLINICAL TRIAL: NCT02340962
Title: Evaluate the Efficacy and Safety of TG-2349 in Combination With Peg-interferon and Ribavirin in Treatment naïve East Asian Subjects With Chronic Hepatitis C Virus Genotype 1b Infection.
Brief Title: Evaluate the Efficacy and Safety of TG-2349 in Subjects With Hepatitis C Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TaiGen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG-2349-03
Record Dates: First submitted 2015-01-08; First posted 2015-01-19 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Experimental): 200 mg TG-2349 (2 capsules) + Interferon or Peg-interferon + Ribavirin
  Interventions: Drug: TG-2349; Drug: Ribavirin; Drug: Interferon Alfa-2a
- Group II (Experimental): 400 mg TG-2349 (4 capsules) + Interferon or Peg-interferon + Ribavirin
  Interventions: Drug: TG-2349; Drug: Ribavirin; Drug: Interferon Alfa-2a

INTERVENTIONS:
Drug: TG-2349 — TG-2349 (Furaprevir) is available as a Swedish orange capsule (size 0) for oral administration. Each capsule contains an equivalent of 100 mg of TG-2349 spray dried solid (SDD) and the following inactive ingredients: microcrystalline cellulose, croscarmellose sodium, sodium lauryl sulfate, magnesium stearate, and colloidal silicon oxide.
Drug: Ribavirin — RBV (Ribavirin or COPEGUS®) is available as a light pink to pink colored, flat, oval-shaped, film-coated tablet for oral administration. Each tablet contains 200 mg of ribavirin and the following inactive ingredients: pregelatinized starch, microcrystalline cellulose, sodium starch glycolate, cornstarch, and magnesium stearate. The coating of the tablet contains Chromatone-P® or Opadry® Pink (made by using hydroxypropyl methyl cellulose, talc, titanium dioxide, synthetic yellow iron oxide, and synthetic red iron oxide), ethyl cellulose (ECD-30), and triacetin.
Drug: Interferon Alfa-2a — IFN (Interferon, Peg-interferon alpha-2a or PEGASYS®) is available as a sterile, preservative-free, colorless to light yellow injectable solution administered subcutaneously.
  Each prefilled syringe of 180 μg/0.5 mL IFN (expressed as the amount of interferon alfa-2a) also contains acetic acid (0.0231 mg), benzyl alcohol (5 mg), polysorbate 80 (0.025 mg), sodium acetate trihydrate (1.3085 mg), and sodium chloride (4 mg) at pH 6 ± 0.5.

SUMMARY:
A Phase 2, Multicenter, Randomized, Open-label, Dose-ranging Study to Evaluate the Efficacy and Safety of TG-2349 in Combination with Peg-interferon and Ribavirin in Treatment Naïve East Asian Subjects with Chronic Hepatitis C Virus Genotype 1b Infection.

DETAILED DESCRIPTION:
It is a multicenter, randomized, open-label study to evaluate the safety, tolerability, and antiviral efficacy of two different doses of TG-2349 combined with Peg-interferon (IFN) and Ribavirin (RBV) in HCV-GT1b treatment naïve East Asian subjects. The treatment duration of TG-2349+IFN+RBV is 12 weeks, with or without an additional 12-week treatment of IFN+RBV, depending on HCV RNA level at On-Treatment Week 4. Approximately 24 subjects will be randomized (1:1) to one of the following 2 treatment groups:

* Group I (n=12): 200 mg TG-2349 (2 capsules) + IFN + RBV
* Group II (n=12): 400 mg TG-2349 (4 capsules) + IFN + RBV Randomization will be stratified by IL28B genotype "CC" or "non-CC". Subjects with HCV RNA < LLOQ (lower limit of quantification), TD (target detected) or TND (target not detected) at Week 4 will receive 12 weeks of TG-2349+IFN+RBV treatment. Subjects with HCV RNA ≥ LLOQ but < 100 IU/mL at Week 4 will receive 12 weeks of TG-2349+IFN+RBV treatment followed by an additional 12 weeks of IFN+RBV treatment. However, subjects with HCV RNA ≥ 100 IU/mL at Week 4 will discontinue the study treatment and complete the Early-Termination (ET) visit. The study will be terminated if 3 or more of the first 12 subjects enrolled across both Groups I and II, or ≥ 25% of subjects thereafter, fail to respond to treatment (i.e., confirmed on-treatment virologic failure or post-treatment relapse). Patients, except those who have achieved SVR12, will be offered the standard of care with Peg-interferon and Ribavirin for duration of 24, 48, or 72 weeks based on Taiwan's regulatory guideline and principal investigator's judgment.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. East Asian subjects, male or female, and age between 18 (or legal adult age) and 70 years, inclusive, at Baseline/Day 1.
3. Body mass index (BMI) in the range of 18.0 to 35.0 kg/m2 (inclusive) and body weight ≥ 40 kg.
4. Presence of chronic hepatitis C (CHC) as documented below:

(1) A positive anti-HCV antibody test or positive HCV RNA or positive HCV genotyping test at least 6 months prior to the Baseline/Day 1 visit or (2) A liver biopsy or FibroTest performed prior to the Baseline/Day 1 visit with evidence of chronic HCV infection, such as the presence of fibrosis and/or inflammation.

5. Positive for anti-HCV antibody at Screening. 6. Presence of an HCV RNA level ≥ 1 x 10000 IU/mL at Screening as determined by the Central Laboratory.

7. Presence of genotype 1b HCV-infection at Screening as determined by the Central Laboratory. Any non-definitive results will exclude the subject from study participation.

8. HCV treatment naïve defined as no prior therapy with any interferon (IFN), ribavirin (RBV), or other approved or investigational HCV-specific agent.

9. Absence of cirrhosis

Cirrhosis as defined as any one of the following:

1. Liver biopsy showing cirrhosis (e.g., Metavir score = 4 or Ishak score ≥ 5).
2. FibroScan showing cirrhosis or results > 12.5 kPa.
3. FibroTest fibrosis score of > 0.58 and APRI (AST: platelet ratio index) of > 2 during Screening.

If no definitive diagnosis of cirrhosis by the above criteria, a liver biopsy is required; liver biopsy results will supersede non-invasive testing results and be considered definitive.

10. Screening ECG without clinically significant abnormalities. 11. Subjects must have the following laboratory parameters at Screening:

1. ALT ≤ 10 × the upper limit of normal (ULN)
2. AST ≤ 10 × ULN
3. Total bilirubin ≤ 1.5 × ULN except history of Gilbert's syndrome. If Gilbert's syndrome is the proposed etiology, the total bilirubin must ≤ 2 × ULN.
4. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
5. Platelet count ≥ 90,000 cells/mm3
6. HbA1c ≤ 8.5%
7. Thyroid stimulating hormone (TSH) and free T4 ≤ ULN
8. Creatinine clearance (CLcr) ≥ 60 mL /min, as calculated by the Cockcroft-Gault equation
9. Serum creatinine ≤ 1.5 × ULN
10. Hemoglobin ≥ 11 g/dL for female subjects; ≥ 12 g/dL for male subjects
11. Albumin ≥ 3.5 g/dL
12. INR (International Normalized Ratio for Prothrombin Time) ≤ 1.5 x ULN unless subject is stable on an anticoagulant regimen affecting INR
13. Anti-nuclear antibodies (ANA) ≤ 1:320. 12. Subject must be of generally good health, with the exception of chronic HCV infection, as determined by Investigator.

13. Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments, including all required Post-Treatment visits.

14. A female subject is eligible to enter the study if it is confirmed that she is:

(1) Not pregnant or nursing. (2) Of non-childbearing potential (i.e., women who have had a hysterectomy, have both ovaries removed or medically documented ovarian failure, or are postmenopausal - women > 50 years of age with cessation (for ≥12 months) of previously occurring menses), or (3) Of childbearing potential (i.e., women who have not had a hysterectomy, have not had both ovaries removed, and have not had medically documented ovarian failure).

Women ≤ 50 years of age with amenorrhea will be considered to be of childbearing potential. These women must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at the Baseline/Day 1 visit prior to randomization. They must also agree to one of the following from Screening until 6 months after the last dose of study drug(s):

- Complete abstinence from intercourse. Periodic abstinence from intercourse (e.g., calendar, ovulation, symptothermal, post-ovulation methods) is not permitted.

Or - Consistent and correct use of 1 of the following methods of birth control listed below, in addition to a male partner who correctly uses a condom, from Screening until 6 months after the last dose of study drug(s):

1. intrauterine device (IUD) with a failure rate of < 1% per year
2. female barrier method: cervical cap or diaphragm with spermicidal agent
3. tubal sterilization
4. vasectomy in male partner
5. hormone-containing contraceptive:

i. implants of levonorgestrel ii. injectable progesterone iii. oral contraceptives (either combined or progesterone only) iv. contraceptive vaginal ring v. transdermal contraceptive patch. 15. Male subjects must agree to consistently and correctly use a condom, while their female partner agrees to use 1 of the methods of birth control listed above, from Screening until 6 months after the last dose of study drug(s).

16. Male subjects must agree to refrain from sperm donation from Screening until at least 6 months after the last dose of study drug(s).

Exclusion Criteria:

1. Presence of cirrhosis.
2. Positive serological test for IgM anti-HAV (hepatitis A virus) antibody or HBsAg at Screening.
3. Positive ELISA test for HIV-1 or HIV-2 at Screening.
4. Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, Wilson disease, alfa-1 antitrypsin deficiency, cholangitis).
5. Donation or loss of more than 400 mL blood within 2 months prior to Baseline/Day 1.
6. Clinically-relevant drug abuse within 12 months of Screening. A positive drug screen will exclude subjects unless it can be explained by a prescribed medication; the diagnosis and prescription must be approved by Investigator.
7. Alcohol misuse as defined by an AUDIT score of ≥ 8.
8. Contraindications to RBV or IFN therapy, including hemoglobinopathies (e.g., thalassemia major or sickle-cell anemia), autoimmune thyroiditis or other autoimmune disorders including autoimmune hepatitis.
9. Pregnant or nursing female or male with pregnant female partner.
10. Use of any prohibited medications within 30 days of the Baseline/Day 1 visit:

(1) Hematologic stimulating agents (e.g., erythropoiesis-stimulating agents [ESAs], granulocyte colony stimulating factor [G-CSF], and thrombopoietin [TPO] mimetics) (2) Chronic use of systemic immunosuppressants including, but not limited to, corticosteroids (prednisone equivalent of > 10 mg/day for > 2 weeks), azathioprine, or monoclonal antibodies (eg, infliximab) (3) Investigational agents or devices for any indication (4) Drugs disallowed per prescribing information of RBV or IFN (5) Any prohibited medications listed in Table 6-2. 11. Known hypersensitivity to RBV, IFN, TG-2349, sulfa drugs, or formulation excipients.

12. Current or prior history of any of the following:

1. Clinically-significant illness (other than HCV) or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol; subjects currently under evaluation for a potentially clinically-significant illness (other than HCV) are also excluded.
2. Gastrointestinal disorder or post operative condition that could interfere with the absorption of the study drugs.
3. Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy.
4. Clinical hepatic decompensation (i.e., ascites, encephalopathy or variceal hemorrhage).
5. Central nervous system (CNS) trauma, seizure disorder, stroke or transient ischemic attack.
6. Solid organ transplantation.
7. Significant cardiac disease (including but not limited to the myocardial infarction based on ECG and/or clinical history).
8. Significant pulmonary disease or porphyria.
9. Clinically significant retinal disease
10. Psychiatric hospitalization, suicide attempt, and/or a period of disability as a result of their psychiatric illness within the last 5 years. Subjects with psychiatric illness (without the prior mentioned conditions) that is well-controlled on a stable treatment regimen for at least 12 months prior to Baseline/Day 1 or has not required medication in the last 12 months may be included.
11. Malignancy within 5 years prior to Screening, with the exception of specific cancers that are entirely cured by surgical resection (basal cell skin cancer, etc). Subjects under evaluation for possible malignancy are not eligible.
12. Significant drug allergy (such as anaphylaxis or hepatotoxicity).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05; Primary Completion 2016-08-12 (Actual); Study Completion 2016-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lung Yu, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- 200 mg TG-2349: 200 mg TG-2349 (2 capsules) + Interferon or Peg-interferon + Ribavirin
- 400 mg TG-2349: 400 mg TG-2349 (4 capsules) + Interferon or Peg-interferon + Ribavirin
Period: Overall Study
Arm/Group | 200 mg TG-2349 | 400 mg TG-2349
Started | 13 | 12
Completed | 12 | 12
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) population includes subjects with genotype 1b HCV infection who were enrolled and received at least one dose of study drugs.
Groups:
- Total: Total of all reporting groups
Arm/Group | 200 mg TG-2349 | 400 mg TG-2349 | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (10.76) | 54.0 (11.91) | 52.3 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 12 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilogram] | 62.8 (13.69) | 64.0 (9.11) | 63.4 (11.49)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Sustained Viral Response at 12 Weeks After the End of Treatment.
Description: Proportion of subjects with HCV RNA< LLOQ (lower limit of quantification), TD (target detected) or TND (target not detected) at 12 weeks after the end of treatment (SVR12) in the Full Analysis Set (FAS) population, which include subjects with genotype 1b HCV infection who were enrolled and received at least one dose of study drugs.
Time Frame: 12 weeks after the end of treatment (SVR12), after 12-week treatments
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 200 mg TG-2349 | 400 mg TG-2349
Number analyzed (Participants) | 13 | 12
Participants | 11 | 10

2. Secondary Outcome: Proportion of Subjects Achieving Sustained Viral Response at 4, 8, and 24 Weeks After the End of Treatment (SVR4, SVR8, and SVR24)
Time Frame: 4, 8, 24 weeks after the end of treatment (SVR4, 8, 24), after 12-week treatments
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 200 mg TG-2349 | 400 mg TG-2349
Number analyzed (Participants) | 13 | 12
Participants
  SVR4 | 12 | 10
  SVR8 | 11 | 10
  SVR24 | 11 | 10

3. Secondary Outcome: Proportion of Subjects Achieving HCV RNA < Lower Limit of Quantification, Target Detected or Target Not Detected (< LLOQ, TD or TND)
Time Frame: The whole treatment period, 12 weeks
Population: Full Analysis Set (FAS) population includes subjects with genotype 1b HCV infection who were enrolled and received at least one dose of study drugs. Missing data were excluded in the dominator of on-treatment visits.
Measure: Count of Participants; unit: Participants
Arm/Group | 200 mg TG-2349 | 400 mg TG-2349
Number analyzed (Participants) | 13 | 12
Participants
  Baseline | 0 | 0
  Day 4 | 1 | 0
  Week 1 | 3 | 4
  Day 10 | 6 | 8
  Week 2 | 9 | 10
  Week 3 | 11 | 10
  Week 4: number analyzed (Participants) | 12 | 12
  Week 4 | 12 | 11
  Week 6: number analyzed (Participants) | 11 | 11
  Week 6 | 11 | 11
  Week 8: number analyzed (Participants) | 11 | 11
  Week 8 | 11 | 11
  Week 10: number analyzed (Participants) | 11 | 11
  Week 10 | 11 | 11
  Week 12: number analyzed (Participants) | 11 | 11
  Week 12 | 11 | 11

4. Secondary Outcome: Proportion of Subjects Achieving HCV RNA < LLOQ, TND
Time Frame: Treatment period (12 to 24 weeks) and after the end of treatment (12 to 24 weeks)
Population: Full Analysis Set (FAS) population includes subjects with genotype 1b HCV infection who were enrolled and received at least one dose of study drugs. Missing data were excluded in the dominator of on-treatment visits, while imputation was performed at post-treatment visits and the dominator for post-treatment visits was the total population.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I | Group II
Number analyzed (Participants) | 13 | 12
Participants
  Baseline | 0 | 0
  Day 4 | 0 | 0
  Week 1 | 1 | 1
  Day 10 | 0 | 3
  Week 2 | 2 | 4
  Week 3 | 4 | 9
  Week 4: number analyzed (Participants) | 12 | 12
  Week 4 | 6 | 9
  Week 6: number analyzed (Participants) | 11 | 11
  Week 6 | 7 | 10
  Week 8: number analyzed (Participants) | 11 | 11
  Week 8 | 11 | 10
  Week 10: number analyzed (Participants) | 11 | 11
  Week 10 | 9 | 11
  Week 12: number analyzed (Participants) | 11 | 11
  Week 12 | 11 | 10
  Post-Treatment Week 4 | 12 | 10
  Post-Treatment Week 8 | 11 | 10
  Post-Treatment Week 12 | 11 | 9
  Post-Treatment Week 24 | 10 | 10

5. Secondary Outcome: Mean Absolute Values in HCV RNA (log10 IU/mL)
Time Frame: Treatment period (12 to 24 weeks) and after the end of treatment (12 to 24 weeks)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | 200 mg TG-2349 | 400 mg TG-2349
Number analyzed (Participants) | 13 | 12
log10 IU/mL
  Baseline | 5.8 (0.83) | 5.9 (0.66)
  Day 4 | 1.9 (0.40) | 2.0 (0.74)
  Week 1 | 1.4 (0.52) | 1.4 (0.54)
  Day 10 | 1.2 (0.19) | 1.1 (0.83)
  Week 2 | 1.0 (0.48) | 1.0 (0.72)
  Week 3 | 0.7 (0.51) | 0.4 (0.78)
  Week 4 | 0.5 (0.54) | 0.4 (0.71)
  Week 6 | 0.4 (0.53) | 0.1 (0.31)
  Week 8 | 0.0 (0.00) | 0.1 (0.31)
  Week 10 | 0.2 (0.42) | 0.0 (0.00)
  Week 12 | 0.0 (0.00) | 0.1 (0.31)
  Post-Treatment Week 4 | 0.0 (0.00) | 0.8 (1.79)
  Post-Treatment Week 8 | 0.2 (0.57) | 0.9 (2.13)
  Post-Treatment Week 12 | 0.5 (1.86) | 1.0 (2.22)
  Post-Treatment Week 24 | 0.1 (0.31) | 0.0 (0.00)

6. Secondary Outcome: Proportion of Subjects Experiencing Virologic Failure During Treatment and Viral Relapse After the End of Treatment.
Time Frame: Treatment period (12 to 24 weeks) and after the end of treatment (12 to 24 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 200 mg TG-2349 | 400 mg TG-2349
Number analyzed (Participants) | 13 | 12
Participants
  Virologic failure | 1 | 2
  On-Treatment failure | 0 | 1
  Post-Treatment relapse | 1 | 1

7. Secondary Outcome: Proportion of Subjects With Abnormal Alanine Aminotransferase (ALT) Levels at Baseline Who Achieved Normal Limit of ALT at Final Treatment Visit.
Time Frame: From baseline (day 1) to the final treatment visit (week 12 or week 24)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 200 mg TG-2349 | 400 mg TG-2349
Number analyzed (Participants) | 13 | 12
Participants
  ALT > ULN at baseline | 7 | 7
  ALT normalization: number analyzed (Participants) | 7 | 7
  ALT normalization | 2 | 5

8. Secondary Outcome: Change From Baseline in HCV RNA (log10 IU/mL)
Time Frame: Treatment period (12 to 24 weeks) and after the end of treatment (12 to 24 weeks)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | 200 mg TG-2349 | 400 mg TG-2349
Number analyzed (Participants) | 13 | 12
log10 IU/mL
  Day 4 | -3.8 (0.51) | -3.9 (0.55)
  Week 1 | -4.4 (0.50) | -4.5 (0.56)
  Day 10 | -4.6 (0.75) | -4.8 (0.78)
  Week 2 | -4.8 (0.91) | -4.9 (1.01)
  Week 3 | -5.0 (1.03) | -5.5 (0.96)
  Week 4 | -5.2 (0.79) | -5.5 (0.73)
  Week 6 | -5.4 (0.86) | -5.7 (0.65)
  Week 8 | -5.8 (0.90) | -5.7 (0.70)
  Week 10 | -5.6 (0.86) | -5.8 (0.67)
  Week 12 | -5.8 (0.90) | -5.7 (0.68)
  Post-Treatment Week 4 | -5.8 (0.86) | -5.1 (1.72)
  Post-Treatment Week 8 | -5.6 (0.88) | -5.0 (2.05)
  Post-Treatment Week 12 | -5.2 (1.81) | -4.8 (2.10)
  Post-Treatment Week 24 | -5.6 (0.83) | -5.8 (0.70)

ADVERSE EVENTS:
Time Frame: through study completion, up to 48 weeks
Arm/Group | Group I | Group II
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/13 | 2/12
Other Adverse Events (participants affected / at risk) | 13/13 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (N=13) | Group II (N=12)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (N=13) | Group II (N=12)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 6 (7)
Neutropenia (Blood and lymphatic system disorders) | 6 (7) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 4 (6) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vesicle (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 5 (5) | 5 (6)
Pyrexia (General disorders) | 2 (2) | 4 (5)
Chest discomfort (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 1 (1) | 1 (1)
Feeling cold (General disorders) | 1 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 1 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (6) | 4 (4)
Headache (Nervous system disorders) | 4 (7) | 3 (3)
Memory impairment (Nervous system disorders) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 3 (3) | 3 (4)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pyuria (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (2)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1) | 1 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Musculoskeletal and connective tissue disorders (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Back pain (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Plantar fasciitis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less